CLINICAL TRIAL: NCT06052605
Title: Healthy Aging in People With Epilepsy Program (HAP-E): Closing the Gap in Epilepsy Care
Brief Title: Healthy Aging in People With Epilepsy Program
Acronym: HAP-E
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Anny Reyes, Postdoctoral Fellow, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAPE2023
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAP-E Epilepsy Participants (Experimental)
  Interventions: Behavioral: Healthy Aging in People with Epilepsy Program

INTERVENTIONS:
Behavioral: Healthy Aging in People with Epilepsy Program — This a 12-week group educational program providing education on healthy aging, chronic disease management, dementia, and modifiable lifestyle dementia risk factors.

SUMMARY:
The goal of this clinical trial is to develop and test an educational program about dementia in older adults living with epilepsy. The main questions it aims to answer are:

1. Can providing education on healthy aging, chronic disease management, dementia, and modifiable lifestyle dementia risk factors improve dementia knowledge and health literacy among older adults with epilepsy?
2. Can aging related education and resources improve quality of life among older adults with epilepsy?

Participants will:

* Complete a 12-week group educational program.
* Complete pre- and post-program evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of epilepsy made by a neurologist, epileptologist, or internist/family medicine physician
* Proficiency in English

Exclusion Criteria:

* Dementia

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Dementia Knowledge | Pre and Post intervention (3 months)
  Dementia Knowledge Assessment Tool was designed to measure change in knowledge of dementia including dementia and its progress, support, and care. It contains 21 true/false items.
Health literacy | Pre and Post intervention (3 months)
  Short Assessment of Health Literacy-English is an 18-item scale assessing adult's ability to read and understand common medical terms.
Health Related Quality of life | Pre and Post intervention (3 months)
  Quality of life in Epilepsy-31 is a self-report questionnaire assessing quality of life in individuals with epilepsy. It measures of overall quality of life, emotional well-being, role limitations due to emotional problems, social support, social isolation, energy/fatigue, worry about seizure, medication effects, health discouragement, work/driving/social function, physical function, pain, role limitations due to physical problems, health perception, and perceived problems with attention/concentration, language, memory.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Califonia, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No